CLINICAL TRIAL: NCT07135765
Title: Paravertebral Muscles Assessment Using High-resolution MRI in Children Suffering From Idiopathic or Neuromuscular Scoliosis
Brief Title: Paravertebral Muscles Assessment Using High-resolution MRI in Idiopathic or Neuromuscular Scoliosis Children
Acronym: MRISCOL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APHP241726; 2024-A02677-40 (Registry Identifier: IDRCB)
Record Dates: First submitted 2025-07-15; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-07

CONDITIONS: Scoliosis; Scoliosis Idiopathic; Scoliosis Neuromuscular
Keywords: scoliosis; MRI; Scoliosis Idiopathic; Scoliosis Neuromuscular; spine; Children
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- idiopathic scoliosis (IS) (Active Comparator)
  Interventions: Procedure: Additional 5 minutes of lying down position during MRI
- neuromuscular scoliosis (NMS) (Active Comparator)
  Interventions: Procedure: Additional 5 minutes of lying down position during MRI

INTERVENTIONS:
Procedure: Additional 5 minutes of lying down position during MRI — During axial MRI for scoliosis assessment, additional 5 minutes of lying down position in order to performing a specific sequence for the study of the vertebral muscles (Diffusion Tensor Imaging).

SUMMARY:
Scoliosis is a common three-dimensional spinal deformity defined by vertebral rotation.

Apart from collapse scoliosis, clinical and radiological similarities have been observed in children with secondary scoliosis of neuromuscular origin and children with idiopathic scoliosis in terms of the location and type of curvature.

It seems relevant to study the axial musculature in these children in more detail, particularly the deep muscles (transversospinales muscles) that have a stabilising and rotational function (multifidi and rotatores).

MRI is a non-invasive, non-irradiating technique used in the aetiological diagnosis of idiopathic scoliosis before adolescence and in the diagnosis of secondary scoliosis. However, the muscles are not specifically studied during these examinations. They are performed to analyse the spinal cord and rule out hinge deformities, although this technique does provide information on the paravertebral muscles.

The muscles of interest should be analysed using the usual sequences, with the addition of a sequence (DTI) specific to the study of deep muscles in children undergoing axial MRI. This adds 5 minutes to the standard MRI procedure.

Several morphological muscle parameters would be thus obtained on specific interest areas and then compared between right and left side and between two groups of children, 5 suffering from idiopathic scoliosis and 5 with neuromuscular scoliosis.

Idiopathic scoliosis corresponds to a heterogeneous group of patients in terms of the location, number and progression of the curves. The research hypothesis is that there may be a subgroup of patients with idiopathic scoliosis whose progression and/or aetiology is muscular in origin.

MRI could then become a routine examination in the assessment of all scoliosis, whether idiopathic or not.

DETAILED DESCRIPTION:
This study is based on the hypothesis that there is a subgroup of patients with idiopathic scoliosis whose onset and/or progression is linked to muscle dysfunction.

This is a prospective, comparative, non-randomised study without a control group, performed in a single centre (Garches Hospital in France is a reference centre for neuromuscular diseases and disabilities). This research is in the field of data collection techniques using imaging methods on two populations of children with scoliosis.

OBJECTIVES The primary objective is the assessment of morphological differences in paravertebral muscles between children with scoliosis of different origins (idiopathic (IS) or neuromuscular (NMS))

Secondary objectives are:

* Assessment of morphological differences between the paravertebral muscles of the convexity and concavity in idiopathic scoliosis
* Assessment of morphological differences between the paravertebral muscles of the convexity and concavity in neuromuscular scoliosis; RESEARCH PROCESS

  1. Selection/Information The selection visit takes place during a routine consultation for the diagnosis/monitoring of scoliosis. Children with idiopathic or neuromuscular scoliosis who, as part of their treatment, need to undergo an axial MRI (spinal cord, pan spinal) and who meet the inclusion criteria could be enrolled.

     Children eligible for the study and their parents, if present, will be offered the opportunity to participate in this study by the investigating physician and will be given the study information sheet.
  2. Inclusion Inclusion is achieved after a minimum reflection period of 48 hours, and no later than the time of the MRI. After obtaining the child's consent and the signature of a parent or guardian, the child will be included in the study.

     They will undergo the MRI scan initially prescribed. If conditions allow, they will be asked to remain still for another 5 minutes while the additional sequence is performed.

     The CAPAS-Q questionnaire (2022 version) will be used to assess physical activity and sedentary behaviour and will be given to the child/adolescent by the investigator to complete. Help will be provided to younger children and children with reading difficulties. The questionnaire will be collected at the end of the visit after it has been completed by the patient.
  3. Data collection and analysis Imaging data will be pseudonymised, collected and analysed with Olea medical Software( olea-medical.com).

Three regions will be defined:

* Region 1 corresponding to the proximal transitional vertebra
* Region 2 corresponding to the apical vertebra (or disc)
* Region 3 corresponding to the distal transitional vertebra These will then be divided into two zones according to the convexity and concavity of the curvature.
* Region 1 convex / Region 1 concave
* Region 2 convex / Region 2 concave
* Region 3 convex / Region 3 concave

Thus, six regions will be defined and seven parameters per region established, i.e. 42 measurements per MRI:

* Cross-sectional area
* Pennation angle
* Number of muscle fibres
* T1 value
* T2 value
* Anisotropy fraction value
* Diffusivity value (average, radial, axial)

Statistical analysis will be descriptive (prospective descriptive study). Quantitative variables will be described by the mean, standard deviation, median and interquartile range.

Qualitative variables will be described by the number of cases and frequency.

Comparisons will be made between the two groups of children with scoliosis according to the aetiology of the scoliosis.

For each of these parameters, non-parametric tests (Wilcoxon, Mann-Whitney) will be performed.

A p-value < 0.05 will be considered significant. No significant difference will be sought between the two groups of children with scoliosis for each parameter, in order to verify the matching of the groups.

* Age
* Gender
* BMI
* CAPAS-Q score (activity and sedentary lifestyle)
* Cobb angle value;

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents aged 10 to 17 years old,
* Scoliosis (idiopathic or neuromuscular) that is not collapsing
* Cobb angle <40°
* Female preferred
* Patient able to walk
* Average or low BMI <20kg/m2
* Signature of informed consent by legal guardians
* Affiliation with a social security scheme (beneficiary or dependent).

Exclusion Criteria:

* Refusal of the patient and/or parents to participate in the study
* Inability to cooperate
* Subject with a contraindication to MRI
* History of spinal surgery
* Not affiliated with a social security scheme (beneficiary or entitled person)

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2025-07-17 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Muscular parameters defined in areas of specific interest and studied in the concavity and convexity of the main curvature: Cross-sectional area | at baseline
  Analysis of differences in several morphological muscle parameters obtained from MRI scans between children with scoliosis (SI versus SNM).
  - Cross-sectional area
  The parameter will be defined in areas of specific interest at the transitional vertebrae and apical vertebrae and will be studied in the concavity and convexity.
Muscular parameters defined in areas of specific interest and studied in the concavity and convexity of the main curvature: Pennation angle | at baseline
  Analysis of differences in several morphological muscle parameters obtained from MRI scans between children with scoliosis (SI versus SNM).
  - Pennation angle
  The parameter will be defined in areas of specific interest at the transitional vertebrae and apical vertebrae and will be studied in the concavity and convexity.
Muscular parameters defined in areas of specific interest and studied in the concavity and convexity of the main curvature: Number of muscle fibres | at baseline
  Analysis of differences in several morphological muscle parameters obtained from MRI scans between children with scoliosis (SI versus SNM).
  - Number of muscle fibres
  The parameter will be defined in areas of specific interest at the transitional vertebrae and apical vertebrae and will be studied in the concavity and convexity.
Muscular parameters defined in areas of specific interest and studied in the concavity and convexity of the main curvature: T1 value | at baseline
  Analysis of differences in several morphological muscle parameters obtained from MRI scans between children with scoliosis (SI versus SNM).
  - T1 value
  The parameter will be defined in areas of specific interest at the transitional vertebrae and apical vertebrae and will be studied in the concavity and convexity.
Muscular parameters defined in areas of specific interest and studied in the concavity and convexity of the main curvature: Anisotropy fraction value | at baseline
  Analysis of differences in several morphological muscle parameters obtained from MRI scans between children with scoliosis (SI versus SNM).
  - Anisotropy fraction value
  These parameters will be defined in areas of specific interest at the transitional vertebrae and apical vertebrae and will be studied in the concavity and convexity.
Muscular parameters defined in areas of specific interest and studied in the concavity and convexity of the main curvature: Diffusivity value | at baseline
  Analysis of differences in several morphological muscle parameters obtained from MRI scans between children with scoliosis (SI versus SNM).
  - Diffusivity value (average, radial, axial)
  These parameters will be defined in areas of specific interest at the transitional vertebrae and apical vertebrae and will be studied in the concavity and convexity.
Muscular parameters defined in areas of specific interest and studied in the concavity and convexity of the main curvature: T2 value | at baseline
  Analysis of differences in several morphological muscle parameters obtained from MRI scans between children with scoliosis (SI versus SNM).
  - T2 value
  These parameters will be defined in areas of specific interest at the transitional vertebrae and apical vertebrae and will be studied in the concavity and convexity.

CONTACTS AND LOCATIONS:
Overall Officials: Hélène Gouz, MD, Principal Investigator — CHU Raymond Poincaré - APHP; Robert Carlier, MD, PhD, Study Director — CHU Raymond Poincaré - APHP
Locations (1):
- CHU Raymond Poincaré - APHP, Garches, France

IPD SHARING:
Plan to Share IPD: Undecided